CLINICAL TRIAL: NCT04390581
Title: A Prospective Study Evaluating the Effectiveness of Juvederm Volift With Lidocaine for Treatment of the Aging Hands
Brief Title: A Study to Evaluate the Effect of Juvederm Volift With Lidocaine on Aging Hands in Participants Age 35 and Older
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-MA-FAS-0628
Record Dates: First submitted 2020-05-07; First posted 2020-05-15 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Skin Depressions; Skin Elasticity; Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Juvéderm® VOLIFT with Lidocaine (Experimental): All participants to be injected with Juvéderm® VOLIFT with Lidocaine in both hands no more than 6ml total per both hands. Optional touch-up will be done on Day 30 according to aesthetic results.
  Interventions: Device: Juvéderm® VOLIFT with Lidocaine

INTERVENTIONS:
Device: Juvéderm® VOLIFT with Lidocaine — Consists of one injection of Juvéderm® VOLIFT with Lidocaine to both hands no more than 6ml for both hands total on Day 1. Optional on Day 30.

SUMMARY:
This study will evaluate the effect of Juvederm Volift with Lidocaine, an injectable gel implant, to treat aging hands of participants 35 and older.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Female and male subjects over 35 years of age
* Has a desire for treatment with hyaluronic acid for skin depressions on both hands
* Must qualify to receive Juvéderm® VOLIFT®™ with Lidocaine as described in the current European Union Juvéderm® VOLIFT®™ with Lidocaine Directions For Use (DFU)
* Accepts the obligation not to receive any other hand cosmetic procedures or treatments at any time during the study (hand creams are permitted)
* Agrees not to change their normal hand care regimen throughout the course of the study.
* Women of childbearing potential must have a negative urine pregnancy test result at baseline (Day 1) and practice a reliable method of contraception throughout the study.

Exclusion Criteria:

* All contraindications as described in the current European Union Juvéderm® VOLIFT®™ with Lidocaine Directions For Use (DFU), as supplied with the product.
* Receiving or planning to receive anticoagulant therapy during the course of the study, or received anticoagulant within 10 days prior to study treatment and 3 days after.
* Receiving or is planning to receive anti-inflammatory drugs (oral/injectable corticosteroids or NSAIDs, e.g., aspirin, ibuprofen), or other substances known to increase coagulation time (vitamins or herbal supplements, e.g., Vitamin E, gingko) for 10 days prior to study treatment and 3 days after
* Undergone hand surgery, tissue grafting, or tissue augmentation with silicone, fat, or other permanent, or semi-permanent dermal fillers or be planning to undergo any of these procedures at any time during the study
* Undergone temporary hand dermal filler injections with any substance within 12 months prior to entry in the study
* Noticeable scarring, active inflammation, infection, cancerous or pre-cancerous lesion, or unhealed wound or have undergone radiation treatment in the area to be treated
* Subject with a dental infection (e.g. infected tooth or paradonitis) or have received dental cleaning within one month of such infection
* Subject with history of hypertrophic scarring on hands
* Any fibrosis or scarring or deformities on the hands - History of neurological disease that may affect peripheral neurological function
* Subjects with a history of Raynaud´s disease or phenomenon, or history of other disease that may affect peripheral circulation
* Subjects with a history of autoimmune disease or joint disease or connective tissue disease (e.g., rheumatoid arthritis, lupus, scleroderma etc.)
* Woman pregnant, lactating, or planning to become pregnant at any time during the study
* Received any investigational product within 30 days prior to study enrollment or be planning to participate in another investigation during the course of this study
* Subject with any skin disease (acute and/or chronic) on the treated zone, likely to interfere with the measured parameters or to put the subject to an undue risk.
* Subject with multiple allergies, anaphylactic shock history, evolutive allergic pathologies.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
At least a 1-point improvement in the Allergan Hand Volume Deficit Scale (AHVDS) by hand from baseline before treatment to 3-month visit. | Month 3
  The Evaluating Investigator will grade each hand using the AHVDS 5-point scale where 0= No visible tendons and veins, 1=No protruding tendons, 2=Protruding tendons, 3=Prominent tendons, 4=Tendons very prominent.

SECONDARY OUTCOMES:
Improvement from baseline to each other post-treatment time points in the Allergan Hand Volume Deficit Scale (AHVDS). | Day 30, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  The Evaluating Investigator will grade each hand using the AHVDS 5-point scale where 0= No visible tendons and veins, 1=No protruding tendons, 2=Protruding tendons, 3=Prominent tendons, 4=Tendons very prominent.
Investigator improvement from baseline to each post-treatment time point using the Global Aesthetic Improvement Scale (GAIS) Investigator | Day 30, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  The Evaluating Investigator will assess the aesthetic improvement of the hands using the GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse.
Subject improvement from baseline to each post-treatment time point using the Global Aesthetic Improvement Scale (GAIS) Subject | Day 30, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  The Subject will assess the aesthetic improvement of the hands using the GAIS 5-point scale where: 2=much improved, 1=improved, 0=no change, -1=worse and -2=much worse.
Change in HAND-Q Hand Appearance Scale from baseline before treatment to each post-treatment timepoint | Day 30, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  The Subjects will answer the HAND-Q Hand Appearance Scale questionnaire before injection (baseline) and at each time points after injection. One questionnaire will be completed globally for both hands, taking into account the worst hand.
Change in skin roughness from baseline before treatment to each post-treatment timepoint using PRIMOS ® 3D Lite for skin roughness measurements | Day 30, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  Measurements of skin microrelief will be performed using PRIMOS ® 3D Lite (Phaseshift Rapid In vivo Measurement Of Skin).
Change in skin moisture from baseline before treatment to each post-treatment timepoint using MoistureMeter D® | Day 30, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  MoistureMeter D® (Delfin Technologies) allows to measure water content of biological tissues
Change in skin elasticity from baseline before treatment to each post-treatment timepoint using Cutometer® | Day 30, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  MPA 580 Cutometer® (Courage & Khazaka) is an in vivo non-invasive method to evaluate skin rheological properties: measures of biological extensibility and elasticity variations. Cutaneous skin elasticity measurement will be performed with a 6mm probe
Injection Site Reactions (ISRs) evaluated by the subject 30 days after each injection using a subject injection site diary. | Day 30
Number of patients experiencing one or more treatment emergent adverse events (TEAEs) | Day 30, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  The number of patients who experienced one more TEAEs
Change in baseline in hand function based on finger goniometer test that will be used to measure any changes in hand function at each post-treatment timepoint. | Day 30, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  A finger goniometer measures range-of-motion (ROM) of finger joints (metacarpophalangeal and interphalangeal). To measure finger flexion and extension.
Change in baseline in hand function based on hand dynamometer test that will be used to measure any changes in hand function at each post-treatment timepoint. | Day 30, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  A hand dynamometer measures the maximum isometric strength of the hand and forearm muscles. The preferred and non-preferred hand is assessed in an alternating sequence until 3 trials had been completed per hand.
Change in baseline in hand function based on pinch gauge test that will be used to measure any changes in hand function at each post-treatment timepoint. | Day 30, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  A pinch gauge is a hand-held medical device that is used for measuring a patient's hand strength. After the first trial score is recorded, the test is repeated with the same instructions for the second and third trials and for the other hand. The scores of three successive trials for each hand tested is averaged.

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (1):
- Eurofins Pharmascan /ID# 233683, Lyon, France

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/